CLINICAL TRIAL: NCT01381185
Title: Phase IV Study of Aspirin and Clopidogrel Therapy Tailored by Functional Thrombocyte Examination (PFA-100, LTA and VerifyNOW) in Acute Myocardial Infarction
Brief Title: REsistance to Aspirin and Clopidogrel in acuTe Myocardial Infarction
Acronym: REACT-MI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FNO-KVO-1; plasek680 (Other: University Hospital Ostrava)
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Acute Myocardial Infarction
Keywords: myocardial infarction; percutaneous coronary intervention (PCI); high platelet reactivity (HPR)
MeSH Terms: conditions — Myocardial Infarction | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard therapy (No Intervention): standard dose of 100mg aspirin qd and 1x75mg Clopidogrel will be given
- ASA/CLP increase (Active Comparator): According to 2 platelet monitoring assays HPR confirmation aspirin will be increased to 200mg qd, clopidogrel to 2x75mg qd
  Interventions: Drug: Aspirin 200mg qd, Clopidogrel 2x75mg qd

INTERVENTIONS:
Drug: Aspirin 200mg qd, Clopidogrel 2x75mg qd — According to 2 platelet monitoring assays HPR confirmation aspirin will be increased to 200mg qd, clopidogrel to 2x75mg qd. This treatment will be given for 30 days from index event (myocardial infarction)
  Other Names: R-130964
  Arms: ASA/CLP increase

SUMMARY:
The purpose of this study is to compare 3 point-of-care methods for monitoring antiplatelet therapy to golden standard (Light transmittance aggregometry-LTA) in high risk population of acute myocardial infarction patients. If two methods (PFA-100, VerifyNOW,Multiplate or LTA) will indicate insufficient antiplatelet blockade/high residual reactivity for aspirin, clopidogrel or both, the dose of aspirin will be increased to 200mg qd and the dose of clopidogrel will be increased to 2x75mg qd.In addition genotyping of CYP2C19 (6 alleles) will be performed.

DETAILED DESCRIPTION:
Dual antiplatelet therapy is the cornerstone of treatment of coronary heart disease after coronary stent implantation. The interindividual response to this therapy is not uniform, however. There are subgroups of patients, where no anticipated antiplatelet effect to either aspirin, clopidogrel or both is reached. The term of aspirin/clopidogrel resistance has been introduced few years ago, most recently it was substituted by more suitable term - high on-treatment residual platelet reactivity (HPR). Although there are many assays to monitor antiplatelet therapy, uncertainty still remains about the correlation of HPR with ischemic vascular events (in-stent thrombosis, myocardial infarction, etc.). Thus platelet aggregation testing is considered to be the most promising method to indicate inappropriate/low response to aspirin/clopidogrel, however the best suited method is not established yet. Up-to date light transmittance aggregometry is widely accepted as golden standard, nonetheless labour intensive and difficult to standardize. On the other hand many point-of-care aggregation testing methods like PFA-100, VerifyNOW, Multiplate etc. have been introduced, their role in clinical practice is uncertain, however. The biggest challenge of today is to determine platelet function assay, which could reliably indicate future ischemic vascular events;moreover it could be potentially used to tailor antiplatelet therapy and precede these events. It was demonstrated, that gene polymorphism - CYP2C19*2 and CYP2C9*3 loss of function is conjugated with an increased occurrence of stent thrombosis. Within the project we also plan to examine 4 alleles which have not been examined in detail before.

ELIGIBILITY:
Inclusion Criteria:

* acute myocardial infarction (verified by troponin I elevation and ST-segment deviation ≥0.1mV in ≥2 contiguous ECG leads persisting for at least 20 minutes and angiographical proof of coronary stenosis )
* preceding antiplatelet medication with aspirin100mg qd/5 and more days before PCI
* pre-treatment with 600mg Clopidogrel loading dose
* preferably patients with drug eluting stent implantation
* signed informed consent

Exclusion Criteria:

* stable/unstable angina pectoris
* active malignancy
* contraindication to antiplatelet therapy
* increased risk of bleeding (trauma, surgery or non-ischemic stroke in last month)
* effective anticoagulation therapy:LMWH, Pradaxa, Xarelto, Warfarin
* known thrombophile disorder
* SIRS
* renal insufficiency (eGFR under 15ml/min)
* severe anemia (<80 g/l)
* polyglobulia (>160 g/l)
* pregnancy
* Hematocrit <0.25 > 0.55

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2011-05; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Platelet inhibition level | 5 days
  The main outcome measure is the difference in platelet inhibition between clopidogrel 1x75mg and 2x75mg in HPR patients

SECONDARY OUTCOMES:
Bleeding Events | 30 days
  TIMI major/minor bleeding Bleeding prediction with Crusade bleeding score (calculator free accessible at http://www.crusadebleedingscore.org/index.html)
Stent thrombosis | 30 days
  In-stent thrombosis will be assessed in 30-days time-frame in all patients included in the trial. -- due to inadequate power of the trial IST cannot be primary outcome measure--

OTHER OUTCOMES:
Ischaemic events (not IST) | 30 days
  unplanned targed vessel revascularisation (TVR), need for coronary - aortic by-pass graft ,myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Jiri Plasek, MD, PhD, Principal Investigator — Department of Cardiology, University Hospital Ostrava; Miroslav Homza, MD, Study Chair — Department of Cardiology, University Hospital Ostrava; Jaromir Gumulec, MD, Study Chair — Institute of clinical Hematology, University Hospital Ostrava
Locations (2):
- Czechia (2):
  - University Hospital Ostrava, Ostrava, Poruba
  - Departement of Laboratory Medicine, Prostejov Hospital, Prostějov

REFERENCES:
- [Background] Marcucci R, Gori AM, Paniccia R, Giusti B, Valente S, Giglioli C, Buonamici P, Antoniucci D, Abbate R, Gensini GF. Cardiovascular death and nonfatal myocardial infarction in acute coronary syndrome patients receiving coronary stenting are predicted by residual platelet reactivity to ADP detected by a point-of-care assay: a 12-month follow-up. Circulation. 2009 Jan 20;119(2):237-42. doi: 10.1161/CIRCULATIONAHA.108.812636. Epub 2008 Dec 31. PMID 19118249
- [Background] Cuisset T, Cayla G, Frere C, Quilici J, Poyet R, Gaborit B, Bali L, Morange PE, Alessi MC, Bonnet JL. Predictive value of post-treatment platelet reactivity for occurrence of post-discharge bleeding after non-ST elevation acute coronary syndrome. Shifting from antiplatelet resistance to bleeding risk assessment? EuroIntervention. 2009 Aug;5(3):325-9. doi: 10.4244/51. PMID 19736156
- [Background] Sibbing D, Byrne RA, Bernlochner I, Kastrati A. High platelet reactivity and clinical outcome - fact and fiction. Thromb Haemost. 2011 Aug;106(2):191-202. doi: 10.1160/TH11-01-0040. Epub 2011 Apr 20. PMID 21505714
- See also: Site info — http://www.fno.cz